CLINICAL TRIAL: NCT03017118
Title: A Randomized Controlled Trial Using Turmeric for Patients With Basal Joint Arthritis
Brief Title: Turmeric for Patients With Basal Joint Arthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Neal Chung-Jen Chen, Medical Doctor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016P001402
Record Dates: First submitted 2016-12-07; First posted 2017-01-11 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Thumb Osteoarthritis
MeSH Terms: interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Turmeric (Experimental): Subjects in this group will receive turmeric (100 mg pastille) 3 times per day for 6 weeks.
  Interventions: Dietary Supplement: Turmeric
- Control (Placebo Comparator): Subjects in this group will receive a placebo pill 3 times per day for 6 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Turmeric — Subjects will receive turmeric (100 mg pastille) 3 times per day for 6 weeks.
  Arms: Turmeric
Other: Placebo — Subjects in the control group will receive a placebo 3 times per day for 6 weeks.
  Arms: Control

SUMMARY:
The aim of this study is to assess whether the use of a commercially available nutraceutical, turmeric, is an effective option to manage pain and stiffness in patients with basal joint arthritis. To conduct a pilot Randomized Controlled Trial evaluating the impact of turmeric on basal joint arthritis.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age or older
* English fluency and literacy
* Seeking care for basal joint pain
* Tender over basal joint
* Positive distraction rotation test (rotation of the thumb metacarpal base while applying axial traction)
* Radiographic evidence of Eaton stage 1 and 2 only

Exclusion Criteria:

* Secondary gains (litigations or worker compensation) procedures that may interfere with patients' motivation for treatment
* Inability or unwillingness to participate in a trial study
* Rheumatoid Arthritis or other inflammatory disorder diagnoses
* Post-traumatic osteoarthritis
* Patients on Coumadin/Steroids/NSAIDs/Tylenol
* Diabetes Mellitus
* Pregnant or lactating women
* Basal joint arthritis of Eaton stage 3
* Patients seeking other treatment for their basal joint arthritis (splint, corticosteroid injection, surgery)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in baseline pain intensity | Enrollment, 6 weeks, and 3 months
  0-10 ordinal rating of pain intensity
Change in baseline disability | Enrollment, 6 weeks, and 3 months
  Disability measured by the QuickDASH

CONTACTS AND LOCATIONS:
Overall Officials: Neal Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States